CLINICAL TRIAL: NCT04966026
Title: Study on the Clinical Characteristics and Outcome of Patients With COPD Combined With Pneumonia
Brief Title: Clinical Characteristics and Outcome of Patients With COPD With Pneumonia
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2017017
Record Dates: First submitted 2021-07-04; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2018-05

CONDITIONS: Pneumonia; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pneumonia; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD combined with CAP inpatients: (1) CAP meets the diagnostic criteria published in our 2016 CAP diagnosis and treatment guidelines; CPOPD and AECOPD meet the diagnostic criteria published in our 2013 COPD diagnosis and treatment guidelines; (2) age ≧ 18 years. Exclusion criteria: (1) age <18 years; (2) pregnancy; (3) positive human immunodeficiency virus (HIV) antibody; (4) suspected or confirmed tuberculosis or fungal infection of the lung.
  Interventions: Other: No inervention

INTERVENTIONS:
Other: No inervention — No inervention

SUMMARY:
To identify the clinical characteristics of patients with chronic obstructive pulmonary disease (COPD) combined with community-acquired pneumonia (CAP) and the factors influencing clinical transition.

DETAILED DESCRIPTION:
To identify the clinical characteristics of patients with chronic obstructive pulmonary disease (COPD) combined with community-acquired pneumonia (CAP) and the factors influencing clinical transition.Compared to other chronic airway diseases, COPD patients can often have CAP in combination, but there is a lack of comparative studies between COPD patients with CAP and non-COPD patients with CAP.

ELIGIBILITY:
Inclusion Criteria:

1. CAP meets the diagnostic criteria published in 2016 Chinese CAP diagnosis and treatment guidelines; CPOPD and AECOPD meet the diagnostic criteria published in Chinese 2013 COPD diagnosis and treatment guidelines;
2. Age ≧ 40years.

Exclusion Criteria:

1. age <40years;
2. pregnancy;
3. positive for human immunodeficiency virus (HIV) antibodies;
4. suspected or confirmed tuberculosis or fungal infection of the lung.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD combined with pneumonia admitted to Peking University Third Hospital from March 1, 2017 to February 28, 2018
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
mortality rate | Day 28 from hospitalization
  mortality rate

SECONDARY OUTCOMES:
Number of days in hospital | through study completion, an average of 1 year
  Number of days in hospital
number of days in ICU | through study completion, an average of 1 year
  number of days in ICU
number of days on mechanical ventilation | through study completion, an average of 1 year
  number of days on mechanical ventilation
cause of using antimicrobial drugs | through study completion, an average of 1 year
  Days of using antimicrobial drugs during hospitalization
hospital fees | through study completion, an average of 1 year
  hospital fees.

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Sun, MD, Principal Investigator — Peking University 3rd Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China